CLINICAL TRIAL: NCT04175223
Title: Study to Measure the Impact of Probiotics on Immune Activation and Neurocognitive Disorders in HIV-positive Patients With Neurocognitive Disorders
Brief Title: Impact of Probiotics in HIV-positive Patients With Neurocognitive Disorders
Acronym: PROCOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-AOI-03
Record Dates: First submitted 2019-09-06; First posted 2019-11-22 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: HIV; Neurocognitive Disorders
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotics (Experimental): probiotic administration
  Interventions: Dietary Supplement: Vivomixx
- without probiotic (No Intervention): no change from the usual care

INTERVENTIONS:
Dietary Supplement: Vivomixx — probiotic administration: administration of two sachets per day (one in the morning and one in the evening) during 6 months
  Arms: probiotics

SUMMARY:
The prevalence of HIV-associated neurocognitive disorders (Human Immunodeficiency Virus) remains high during the era of effective triple therapy. The main clinical phenotypes of cognitive impairment are currently represented by asymptomatic neurocognitive neurocognitive impairment (ANI) and mild neurocognitive disorders (MND). In contrast, HIV-associated dementia has almost disappeared.

Among the hypotheses to explain the persistence of such a high prevalence is the persistent activation of the immune system despite virological success. This chronic immune activation is believed to be responsible for an inflammatory response and therefore for accelerated cell aging. Several organ complications in HIV-positive patients have been associated with high markers of immune activation.

Among the causes of chronic immune activation in virologically controlled patients, an imbalance in the intestinal flora is suspected. In fact, shortly after HIV infection, the virus causes significant apoptosis of intestinal lymphocytes, responsible for a loss of integrity of the intestinal barrier and an imbalance of flora, defined as "dysbiosis".

Loss of epithelial integrity and intestinal dysbiosis are suspected of causing systemic passage of bacterial fragments, of which lypopolisaccharide is best known, resulting in chronic activation of the immune system. Several studies suggest a link between digestive bacterial translocation and HIV-related neurocognitive disorders. An improvement in intestinal dysbiosis could therefore contribute to reducing immune activation and the severity of cognitive impairment. A recent study showed that probiotics can reduce levels of neopterin, a marker of monocytic activation, in the cerebrospinal fluid of HIV-positive patients without neurological symptoms.

Our objective is to evaluate the impact of probiotic supplementation on immune activation and cognitive performance in virologically controlled HIV-positive patients with a diagnosis of ANI or MND. The potential improvement of cognition through probiotic treatment could therefore improve their quality of life at a lower cost than a drug and without the risk of serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed informed consent
* Patients infected with HIV-1
* Patients with undetectable viral load and stable antiretroviral therapy for at least 6 months
* Patients with HIV-related neurocognitive disorders of the ANI or MND type, to be confirmed by neuropsychological assessment at inclusion
* Outpatient patients, over 18 years of age
* Patients with social security coverage

Exclusion Criteria:

* Patients infected with HIV-2
* Patients who have not been on stable antiretroviral therapy and have been virologically successful for at least 6 months
* Patients who have been treated during the primary infection phase, taking into account the potential risks of impact on intestinal lymphocyte apoptosis and therefore on the microbiota
* Patients who do not have HIV-related neurocognitive disorders such as ANI or MND
* Patients refusing to participate in the study
* Patients consuming probiotics at inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
measurement of the immune activation and Serum inflammation markers | 6 months
  The immune activation is composed with the following elements (quantity of serum immune activation and inflammation markers : sCD14 (ng/mL), sCD163 (ng/mL), TNF-alpha (ng/ml) , IL-1 (ng/ml) , IL-6 (ng/ml) , IL-8 (ng/ml) , D-Dimeres (ng/ml), hCRP (ng/ml), MCP-1(ng/ml), IP-10 (ng/ml), Neurofilaments light chain (log10 ng/ml) and Lipopolysaccharide (ng/ml)) , at inclusion and after 6 months of probiotic supplementation in the 2 groups wwith laboratory tests.
  The immune activation is the result of the multiple measurements. there is no units of measure and it's not an aggregation of the measurement.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CH Cannes, Cannes
  - CHU Montpellier, Montpellier
  - CHU de Nice, Nice